CLINICAL TRIAL: NCT01407588
Title: Manual Compared to Magnetic Navigation in Ablation for Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); SINTEF Health Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2010/3345-2
Record Dates: First submitted 2011-06-08; First posted 2011-08-02 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2017-03

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Magnetic navigation (Experimental)
  Interventions: Procedure: Magnetic navigation
- Manual navigation (Experimental)
  Interventions: Procedure: Ablation performed with manual navigation

INTERVENTIONS:
Procedure: Magnetic navigation — Ablation with use of the magnetic navigation system
  Arms: Magnetic navigation
Procedure: Ablation performed with manual navigation — Atrial fibrillation ablation performed with manual navigation
  Arms: Manual navigation

SUMMARY:
The purpose of this study is to compare manual and magnetic navigation in ablation for atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing ablation for atrial fibrillation at St. Olavs Hospital
* Implanted Reveal

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Number of participants with recurrence of atrial fibrillation after ablation | 2 years
  If the patient have had recurrence or not of atrial fibrillation after ablation. An implanted arrhythmia loop recorder (Reveal XT) is used for monitoring. Recurrence is defined as an attack of atrial fibrillation of more than 2 minutes. It will also be specified if the patient is referred for a second ablation procedure.

SECONDARY OUTCOMES:
Procedure time | Day 1(after ablation procedure)
  Duration of the ablation procedure
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Day 1(after ablation procedure)
  Complications during and after the ablation procedure. Major: pericardial tamponade, permanent atrioventricular (AV) block, major bleeding, cerebral embolus, infection, heart failure, death. Minor: minor bleeding and temporary AV block.
Exposure of radiation to health personnel involved in the procedure | Day 1(after ablation procedure)
  Total time with use of of radiation equipment. Radiation exposure of the operator.
Amount of analgetics and sedatives given during procedure | Day 1
  As a measure of pain and discomfort experienced by the patient during the procedure, the amount of medications are assessed
Pain | After ablation(day 1)
  Pain scores on the Visual Analog Scale
Numbers of and types of catheters used | During ablation(Day1)
  As a measure of resources needed for the procedure, the catheters used are registered. Numbers of and type of catheters are registered and total cost calculated.
Time with active ablation | During the procedure(Day 1)
  Total time that electrical current has been used during the ablation
Total time nurses are occupied with the ablation | During the ablation(day 1)
  As a measure of cost and resources needed for the procedure
Myocardial damage | After ablation(day 1)
  Measured by Troponin-t and CK-MBAs
Cardiac volumes and function | 1 year
  Measured by echocardiography
Quality of life | 2 years
  Measured by SF-36 and atrial fibrillation symptoms and severity checklist

CONTACTS AND LOCATIONS:
Overall Officials: Jan Paal Loennechen, PhD, Study Chair — St. Olavs Hospital
Locations (1):
- Norwegian University of Science and Technology, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No